CLINICAL TRIAL: NCT01989520
Title: An Open-label, Single Centre Relative Bioavailability Study With an Adaptive Design Comparing up to 5 Solid Oral AZD5069 Formulations After Single Dose Administration to Healthy Volunteers
Brief Title: Study to Investigate Relative Bioavailability of up to Five Different Formulations of AZD5069
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D3551C00002
Record Dates: First submitted 2013-11-15; First posted 2013-11-21 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Uncontrolled and Persistent Asthma
Keywords: Relative bioavailability, Healthy volunteers, Neutrophils

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Treatment A (Experimental): Phase IIb formulation
  Interventions: Drug: Phase IIb formulation
- Treatment B (Experimental): Putative phase III formulation
  Interventions: Drug: Putative phase III formulation
- Treatment C (Experimental): Slow dissolution variant 1
  Interventions: Drug: Slow dissolution variant 1
- Treatment D (Experimental): Slow dissolution variant 2
  Interventions: Drug: Slow dissolution variant 2
- Treatment E (Experimental): Optional treatment that may use one of 3 45 mg (intermediate dissolution variant) of AZD5069
  Interventions: Drug: Test treatment E

INTERVENTIONS:
Drug: Phase IIb formulation — Single oral dose 45mg AZD5069
  Arms: Treatment A
Drug: Putative phase III formulation — Single oral dose 45mg AZD5069
  Arms: Treatment B
Drug: Slow dissolution variant 1 — Single oral dose 45mg AZD5069
  Arms: Treatment C
Drug: Slow dissolution variant 2 — Single oral dose 45mg AZD 5069
  Arms: Treatment D
Drug: Test treatment E — Tablet formulation E, 45 mg (intermediate dissolution variant) of AZD5069
  Arms: Treatment E

SUMMARY:
Study to investigate relative bioavailability of up to five different formulations of AZD5069

DETAILED DESCRIPTION:
An Open-label, Single Centre Relative Bioavailability Study With an Adaptive Design Comparing up to 5 Solid Oral AZD5069 Formulations After Single Dose Administration to Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and/or female volunteers aged 18 to 50 years (inclusive).
2. Non-smokers or ex-smokers with no smoking history for the last 3 months prior to screening.
3. Body mass index (BMI) ≥18.0 and ≤30.0 kg/m2 calculated from height and weight at screening; minimum (min) weight 50 kg and maximum (max) weight 100 kg.
4. Healthy volunteers with neutrophil counts within the laboratory range at screening.

   -

Exclusion Criteria:

1. A definite or suspected personal history of severe allergy, intolerance or hypersensitivity or ongoing allergy to drugs with a similar chemical structure or class to AZD5069 and/or the excipients, as judged to be clinically relevant by the Investigator.
2. Healthy volunteers who have previously received AZD5069.
3. Volunteers with latent tuberculosis as suggested by their history and judged by the Investigator; confirmatory testing with eg, Quantiferon(R) -TB Gold may be done if required.
4. Volunteers who have received live or live-attenuated vaccine in the 2 weeks prior to the first administration of the IP -

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2014-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Description of pharmacokinetics of AZD5069 and its metabolite in terms of area under plasma concentration-time curve from time zero to the time of last quantifiable analyte concentration and extrapolated to infinity (AUC(0-last) and AUC) | Samples taken predose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, and 24 hours postdose
  Curve taken during each of the 5 treatments
Description of pharmacokinetics of AZD5069 and its metabolite in terms of observed maximum plasma concentration (Cmax), plasma concentration measured at 12 hours (C12h), Cmax/C12h ratio, Cmax/AUC ratio, terminal rate constant (λz) | Sample taken predose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, and 24 hours postdose
  Curve taken during each of the 5 treatments
Description of pharmacokinetics of AZD5069 and its metabolite in terms of terminal half-life (t½λz), time to reach maximum plasma concentration (tmax) | Sample taken predose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, and 24 hours postdose
  Curve taken during each of the 5 treatments
Description of pharmacokinetics of AZD5069 and its metabolite in terms of apparent systemic clearance (CL/F) (AZD5069 only), and apparent volume of distribution (Vz/F) (AZD5069 only) | Sample taken predose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, and 24 hours postdose
  Curve taken during each of the 5 treatments

SECONDARY OUTCOMES:
Description of effect on neutrophils in terms of circulating neutrophil numbers reported as absolute circulating neutrophil counts (ANC). The minimum absolute neutrophil count (ANCmin) and the time to ANCmin (ANCtmin) | Baseline sample taken at predose day 1 and then 2, 4, 6, 8, 10, 12, and 24 hours postdose
  Samples taken during each of the 5 treatments
Description of effect on neutrophils in terms of mean of ANC values from predose to 24 hours postdose (ANCmean), the minimum of the ANC ratio values (ANCmin,ratio) | Baseline sample taken at predose day 1 and then 2, 4, 6, 8, 10, 12, and 24 hours postdose
  Samples taken during each of the 5 treatments
Description of effect on neutrophils in terms of the mean of ANC ratio values calculated baseline to 24 hours post dose (ANCmean,ratio) | Baseline sample taken at predose day 1 and then 2, 4, 6, 8, 10, 12, and 24 hours postdose
  Samples taken during each of the 5 treatments

CONTACTS AND LOCATIONS:
Overall Officials: Olufeyikemi Oluwayi, MD, Principal Investigator — Quintiles London UK; Bengt Larssons, MD, Study Director — Astrazeneca Mölndal, Sweden
Locations (1):
- Research Site, London, United Kingdom

REFERENCES:
- [Derived] Cullberg M, Arfvidsson C, Larsson B, Malmgren A, Mitchell P, Wahlby Hamren U, Wray H. Pharmacokinetics of the Oral Selective CXCR2 Antagonist AZD5069: A Summary of Eight Phase I Studies in Healthy Volunteers. Drugs R D. 2018 Jun;18(2):149-159. doi: 10.1007/s40268-018-0236-x. PMID 29856004
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1889&filename=D3551C00002_Study_Synopsis.pdf